CLINICAL TRIAL: NCT02544620
Title: Out Patient Surgery for Total Knee and Hip Replacement and Unicompartmental Knee Replacement - a Feasibility Study
Status: Completed | Type: Observational
Sponsor: Kirill Gromov (Other)
Collaborators: Rigshospitalet, Denmark (Other); Vejle Hospital (Other); Holsterbro Sygehus, DK (Unknown)
Responsible Party: Sponsor-Investigator, Kirill Gromov, MD, PhD, Hvidovre University Hospital
Organization: Hvidovre University Hospital (Other)
Other Study IDs: HVH-SK-TKA-THA-UKA
Record Dates: First submitted 2015-09-06; First posted 2015-09-09 (Estimated); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Total Hip arthroplasty: * Unselected primary THA
  * American Society of Anesthesiologists (ASA) score I/II
  * Can be operated as #1 or #2
  * No sleep apnea treated with Continuous positive airway pressure (CPAP)
  Interventions: Other: Does fulfil of discharge criteria on the day of the surgery; Other: Does not fulfil of discharge criteria on the day of the surgery
- Total Knee arthroplasty: * Unselected primary TKA
  * American Society of Anesthesiologists (ASA) score I/II
  * Can be operated as #1 or #2
  * No sleep apnea treated with Continuous positive airway pressure (CPAP)
  Interventions: Other: Does fulfil of discharge criteria on the day of the surgery; Other: Does not fulfil of discharge criteria on the day of the surgery
- unicompartmental knee arthroplasty: * Unselected primary UKA
  * American Society of Anesthesiologists (ASA) score I/II
  * Can be operated as #1 or #2
  * No sleep apnea treated with Continuous positive airway pressure (CPAP)
  Interventions: Other: Does fulfil of discharge criteria on the day of the surgery; Other: Does not fulfil of discharge criteria on the day of the surgery

INTERVENTIONS:
Other: Does fulfil of discharge criteria on the day of the surgery
Other: Does not fulfil of discharge criteria on the day of the surgery

SUMMARY:
The purpose of this study is to evaluate feasibly of outpatient Total Knee Replacement, Total Hip Replacement and Unicompartmental Knee Replacement in a modern fast-track setup. The design is as an observational prospective study, evaluating patients that fulfil discharge criteria on the day of the surgery. The investigators will further evaluate safety aspects, such a early morbidity and mortality, as well as patient satisfaction.

DETAILED DESCRIPTION:
Fast-track total hip arthroplasty (THA), total knee arthroplasty (TKA) and Unicompartmental Knee arthroplasty (UKA) with length of stay (LOS) of 1-3 is a well established concept for treating hip and knee osteoarthritis, resulting in short reconvalescence, high patient satisfaction, and an excellent safety profile (lower or similar mortality / morbidity compared to conventional pathways with longer LOS). LOS have been significantly reduced during the past decade, and several centers have published even shorter hospitals stays: <24 hours, with patients staying the night at the hospital but also outpatient surgery, with patients being discharged on the day of surgery.

However, these proposed pathways with extremely short LOS, are performed on very selected patients, with few details on patient satisfaction, outcome and most important patient safety. Therefore, it is not possible to draw conclusions on feasibility of outpatient THA, TKA and UKA surgery in a general and unselected population. Further on, there is a need for investigation of safety aspects of outpatient surgery in respect to mortality, morbidity, patient satisfaction and patient reported outcomes. As some, most likely healthy and younger, patients might benefit from outpatient surgery - eg discharge on the day of surgery, while others might not; the first step is to identify the patients that are suitable for outpatient THA and TKA surgery and investigate the safety aspects in respect to mortality, morbidity, patient satisfaction and patient reported outcomes.

Aim:

The aim of this study is to investigate "feasibility" and "safety" of outpatient THA, TKA and UKA surgery, respectively as follows:

Feasibility

* Proportion of patients, that can be included in the study according to inclusion criteria stated below, and be evaluated for potential same-day discharge (I) (I = included)
* Proportion of included patients (I), that are discharged on the day of surgery (U) and those who are not discharged and stay for >1 day (B)
* Identify reasons for patients not being able to be discharged on the day of surgery (B)

Safety

* risk for complications (morbidity) in group (U) compared to group (B) (are there complications that potentially could have been avoided is the patient was not discharged)
* readmissions in group (U ) compared to group (B) within 90 days
* mortality in group (U ) compared to group (B) within 90 days
* patient satisfaction in group (U ) compared to group (B)
* Patient reported outcome (Oxford knee score + range of motion for TKA and UKA group, and Oxford hip score for THA group) in group (U) compared to group (B)
* contacts to primary sector in group (U ) compared to group (B) within 7 days.
* use of rescue morphine (pain journal) for 7 days post op in group (U ) compared to group (B)

ELIGIBILITY:
Inclusion Criteria:

* Unselected primary THA/TKA
* ASA score I/II
* Can be operated as #1 or #2
* No sleep apnea treated with CPAP

Exclusion Criteria:

* Selected primary THA/TKA
* ASA score > 2
* Cannot be operated as #1 or #2
* Sleep apnea treated with CPAP

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Unselected primary THA/TKA/UKA
  * ASA score I/II
  * Can be operated as #1 or #2
  * No sleep apnea treated with CPAP
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2015-09; Primary Completion 2018-08-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Fulfilment of same day discharge criteria | 12 hours
  On the days of surgery following discharge criteria are continuously evaluated:
  * < 500 ml intraoperative blood loss
  * Back in patient ward <15.00
  * Received instruction from physiotherapist and is safely mobilized
  * No clinical symptoms of anemia
  * Pain <3 while resting, <5 during exercise.
  * Spontaneous urination
  * Post op x-ray is performed and approved
  * Relatives or friends with patient for >24 hours
  * Motivated and accepts same day discharge
  * Standard discharge criteria fulfilled
  * Can be discharged before 20.00
  If all of the above criteria are fulfilled, the patient can be discharged

SECONDARY OUTCOMES:
Readmissions | 3 months
Patient reported satisfaction | 3 months
  OKS (Oxford Knee score) and ROM (Range og motion) for TKA and UKA, OHS for THA
Use of rescue morphine | 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Hvidovre Hospital, Hvidovre, Denmark